CLINICAL TRIAL: NCT02778113
Title: A Single Site, Randomized, Four-Way, Four-Period PK/PD Crossover Phase 1 Clinical Study in 16 Fasted Healthy Adult Volunteers Receiving 3 Dose Levels of Intranasally Administered Glucagon and One Dose Level of Glucagon Administered by Subcutaneous Injection
Brief Title: A Study of Glucagon Administered in Different Forms and Routes to Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Locemia Solutions ULC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 16424; I8R-MC-IGBD (Other: Eli Lilly and Company); AMG 101 (Other: AMG Medical Inc.); GUO-P1-557 (Other: AMG Medical Inc.)
Record Dates: First submitted 2016-05-18; First posted 2016-05-19 (Estimated); Results first posted 2019-09-19 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2016-05

CONDITIONS: Healthy
MeSH Terms: interventions — Glucagon

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Nasal Glucagon (NG) - 0.5 mg (Experimental): Ng dose at 0.5 milligram (mg) administered once in one of four study periods.
  Interventions: Drug: Nasal Glucagon
- NG - 1.0 mg (Experimental): Ng dose at 1.0 milligram (mg) administered once in one of four study periods.
  Interventions: Drug: Nasal Glucagon
- NG - 2.0 mg (Experimental): Ng dose at 2.0 milligram (mg) administered once in one of four study periods.
  Interventions: Drug: Nasal Glucagon
- SC Glucagon 1 mg (Active Comparator): Subcutaneous (SC) glucagon dose of 1 mg, in one of four study periods.
  Interventions: Drug: Glucagon

INTERVENTIONS:
Drug: Nasal Glucagon — Administered intranasally.
  Other Names: AMG 504-1; LY900018
  Arms: NG - 1.0 mg; NG - 2.0 mg; Nasal Glucagon (NG) - 0.5 mg
Drug: Glucagon — Administered SC.
  Arms: SC Glucagon 1 mg

SUMMARY:
The main purpose of this study was to evaluate the safety and tolerability of nasal glucagon (NG). The study drug was delivered into the participant's nostril (intranasally) or was given as an injection just under the skin (subcutaneously) once in each of four study periods. The study lasted about 23 days for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) greater than or equal to 20.00 and below or equal to 28.00 kg/m².
* Light-, non- or ex-smokers.
* Have no clinically significant diseases captured in the medical history or evidence of clinically significant findings on physical examination and/or clinical laboratory evaluations (hematology, biochemistry, ECG and urinalysis).

Exclusion Criteria:

* Presence of any nose piercings.
* History of significant hypersensitivity to glucagon or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs.
* Presence of significant gastrointestinal, liver or kidney disease, or any other conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs or known to potentiate or predispose to undesired effects.
* Presence of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic or dermatologic disease.
* Presence of clinically significant findings on nasal examination and bilateral anterior rhinoscopy.
* Fasting blood glucose above 5.0 millimoles per liter (mmol/L) at screening, following a 12-hour fasting period.
* Fasting blood glucose assessed with a glucose meter above 5.5 mmol/L 0.5 hour before each dosing.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2011-10; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mount Royal, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a four-period crossover study in which participants received a single dose of study drug in each period, with seven days between each dose.
Groups:
- Sequence 1 (T1/T2/T3/T4): Treatment (T1) = nasal glucagon (NG) dose of 0.5 milligram (mg), T2 = NG dose of 1 mg, T3 = NG dose of 2 mg, T4 = subcutaneous (SC) glucagon dose of 1 mg. In each of four study periods, a single dose of NG was administered or SC glucagon was administered.
- Sequence 2 (T2/T3/T4/T1): T2 = NG dose of 1 mg, T3 = NG dose of 2 mg, T4 = SC glucagon dose of 1 mg, T1 = NG dose of 0.5 mg. In each of four study periods, a single dose of NG was administered or SC glucagon was administered.
- Sequence 3 (T3/T4/T1/T2): T3 = NG dose of 2 mg, T4 = SC glucagon dose of 1 mg, T1 = NG dose of 0.5 mg, T2 = NG dose of 1 mg. In each of four study periods, a single dose of NG was administered or SC glucagon was administered.
- Sequence 4 (T4/T1/T2/T3): T4 = SC glucagon dose of 1 mg, T1 = NG dose of 0.5 mg, T2 = NG dose of 1 mg, T3 = NG dose of 2 mg. In each of four study periods, a single dose of NG was administered or SC glucagon was administered.
Period: Study Period One
Arm/Group | Sequence 1 (T1/T2/T3/T4) | Sequence 2 (T2/T3/T4/T1) | Sequence 3 (T3/T4/T1/T2) | Sequence 4 (T4/T1/T2/T3)
Started | 4 | 4 | 4 | 4
Received Study Drug | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Study Period Two
Arm/Group | Sequence 1 (T1/T2/T3/T4) | Sequence 2 (T2/T3/T4/T1) | Sequence 3 (T3/T4/T1/T2) | Sequence 4 (T4/T1/T2/T3)
Started | 4 | 4 | 4 | 4
Received Study Drug | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Study Period Three
Arm/Group | Sequence 1 (T1/T2/T3/T4) | Sequence 2 (T2/T3/T4/T1) | Sequence 3 (T3/T4/T1/T2) | Sequence 4 (T4/T1/T2/T3)
Started | 4 | 4 | 3 (One participant completed study period two, but did not enter study period three.) | 4
Received Study Drug | 4 | 4 | 3 | 4
Completed | 4 | 4 | 3 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Study Period Four
Arm/Group | Sequence 1 (T1/T2/T3/T4) | Sequence 2 (T2/T3/T4/T1) | Sequence 3 (T3/T4/T1/T2) | Sequence 4 (T4/T1/T2/T3)
Started | 3 (One participant completed study period three, but did not enter study period four.) | 4 | 2 (One participant completed study period three, but did not enter study period four.) | 4
Received Study Drug | 3 | 4 | 2 | 4
Completed | 3 | 4 | 2 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- All Participants: In each of four study periods, a single dose of either NG or SC glucagon was administered.
Arm/Group | All Participants
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 14
  Black | 1
  Other | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs)
Description: Safety and tolerability evaluated through the assessment of adverse events. A SAE (serious adverse event) was defined as any untoward medical occurrence in a clinical investigation, which did not necessarily have a causal relationship with this treatment.
  A summary of other non-serious AEs, and all SAE's, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Baseline through Study Completion (Day 23)
Population: All randomized participants who entered study period four.
Measure: Count of Participants; unit: Participants
Groups:
- NG 0.5 mg: Nasal glucagon (NG) dose of 0.5 milligram (mg).
- NG 1 mg: NG dose of 1 mg.
- NG 2 mg: NG dose of 2 mg.
- SC Glucagon 1 mg: Subcutaneous (SC) glucagon dose of 1 mg.
Arm/Group | NG 0.5 mg | NG 1 mg | NG 2 mg | SC Glucagon 1 mg
Number analyzed (Participants) | 15 | 14 | 16 | 15
Participants | 0 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Time Zero to T (AUC[0-tlast]) of Baseline Adjusted Glucagon
Time Frame: Day 1: -0.5, -0.25, 0, 0.08, 0.17, 0.25, 0.33, 0.5, 0.67, 1.0, 1.5, 2, 2.5, 3 and 4 hours post dose for each treatment
Population: All randomized participants with evaluable PK data. In the NG 0.5 mg arm, all participants had serum glucagon levels that were below the lower limit of quantification (100 picogram per milliliter [pg/mL]) except for one participant at one time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picogram*hour per milliliter (pg*h/mL)
Groups:
- NG 0.5 mg: NG dose of 0.5 mg.
- SC Glucagon 1 mg: SC glucagon dose of 1 mg.
Arm/Group | NG 0.5 mg | NG 1 mg | NG 2 mg | SC Glucagon 1 mg
Number analyzed (Participants) | 1 | 7 | 15 | 15
picogram*hour per milliliter (pg*h/mL) | NA (NA) — n=1. Individual value was 4.42 pg*h/ml. | 38.9 (483) | 293 (172) | 2060 (68)

3. Secondary Outcome: PK: Area Under the Curve Extrapolated to Infinity (AUC[0-inf]) of Baseline Adjusted Glucagon
Time Frame: Day 1: -0.5, -0.25, 0, 0.08, 0.17, 0.25, 0.33, 0.5, 0.67, 1.0, 1.5, 2, 2.5, 3 and 4 hours post dose for each treatment
Population: All randomized participants with evaluable PK data. AUC(0-inf) could not be calculated for the NG 0.5 mg arm, because all participants had serum glucagon levels below the lower limit of quantification (100 pg/mL) except for one participant at one time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Arm/Group | NG 0.5 mg | NG 1 mg | NG 2 mg | SC Glucagon 1 mg
Number analyzed (Participants) | 0 | 1 | 5 | 14
pg*h/mL |  | NA (NA) — n=1. Individual value was 323 pg*h/mL. | 589 (50) | 2250 (66)

4. Secondary Outcome: PK: Time to Maximum Concentration (Tmax) of Baseline Adjusted Glucagon
Time Frame: Day 1: -0.5, -0.25, 0, 0.08, 0.17, 0.25, 0.33, 0.5, 0.67, 1.0, 1.5, 2, 2.5, 3 and 4 hours post dose for each treatment
Population: All randomized participants with evaluable PK data. In the NG 0.5 mg arm, all participants had serum glucagon levels that were below the lower limit of quantification (100 pg/mL) except for one participant at one time point.
Measure: Median (Full Range); unit: hour (h)
Arm/Group | NG 0.5 mg | NG 1 mg | NG 2 mg | SC Glucagon 1 mg
Number analyzed (Participants) | 1 | 7 | 15 | 15
hour (h) | 0.17 [0.17 to 0.17] | 0.25 [0.17 to 0.28] | 0.25 [0.17 to 0.67] | 0.33 [0.11 to 0.67]

5. Secondary Outcome: PK: Maximum Change From Baseline Concentration (Cmax) of Glucagon
Time Frame: Day 1: -0.5, -0.25, 0, 0.08, 0.17, 0.25, 0.33, 0.5, 0.67, 1.0, 1.5, 2, 2.5, 3 and 4 hours post dose for each treatment
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picogram per milliliter (pg/mL)
Arm/Group | NG 0.5 mg | NG 1 mg | NG 2 mg | SC Glucagon 1 mg
Number analyzed (Participants) | 1 | 7 | 15 | 15
picogram per milliliter (pg/mL) | NA (NA) — n=1. Individual value was 52.0 pg/mL. | 217 (231) | 1000 (104) | 3260 (59)

6. Secondary Outcome: Pharmacodynamics (PD): Area Under the Effect Concentration Time Curve (AUEC₀-₄) of Glucose
Time Frame: Day 1: -0.5, -0.25, 0, 0.08, 0.17, 0.25, 0.33, 0.5, 0.67, 1.0, 1.5, 2, 2.5, 3 and 4 hours post dose for each treatment
Population: All randomized participants with evaluable PD data.
Measure: Mean (Standard Error); unit: millimole*hour per liter (mmol*h/L)
Arm/Group | NG 0.5 mg | NG 1 mg | NG 2 mg | SC Glucagon 1 mg
Number analyzed (Participants) | 15 | 14 | 16 | 15
millimole*hour per liter (mmol*h/L) | -0.168 (0.202) | 0.0617 (0.177) | 0.566 (0.324) | 0.448 (0.490)

7. Secondary Outcome: PD: Time to Maximum Concentration (Tmax) of Baseline-Adjusted Glucose
Time Frame: Day 1: -0.5, -0.25, 0, 0.08, 0.17, 0.25, 0.33, 0.5, 0.67, 1.0, 1.5, 2, 2.5, 3 and 4 hours post dose for each treatment
Population: All randomized participants with evaluable PD data.
Measure: Median (Full Range); unit: hour (h)
Arm/Group | NG 0.5 mg | NG 1 mg | NG 2 mg | SC Glucagon 1 mg
Number analyzed (Participants) | 15 | 14 | 16 | 15
hour (h) | 0.33 [0.17 to 0.67] | 0.36 [0.25 to 0.50] | 0.50 [0.33 to 0.67] | 0.37 [0.25 to 0.67]

8. Secondary Outcome: PD: Baseline-Adjusted Glucose Maximum Concentration (BGmax)
Time Frame: Day 1: -0.5, -0.25, 0, 0.08, 0.17, 0.25, 0.33, 0.5, 0.67, 1.0, 1.5, 2, 2.5, 3 and 4 hours post dose for each treatment
Population: All randomized participants with evaluable PD data.
Measure: Mean (Standard Error); unit: millimole per liter (mmol/L)
Arm/Group | NG 0.5 mg | NG 1 mg | NG 2 mg | SC Glucagon 1 mg
Number analyzed (Participants) | 15 | 14 | 16 | 15
millimole per liter (mmol/L) | 0.811 (0.119) | 1.92 (0.173) | 3.20 (0.252) | 3.28 (0.326)

ADVERSE EVENTS:
Time Frame: First dose of study drug (Day 1) until post-study completion (Day 23)
Description: All randomized participants who entered study period four.
Arm/Group | NG 0.5 mg | NG 1 mg | NG 2 mg | SC Glucagon 1 mg
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14 | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 2/15 | 6/14 | 8/16 | 6/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NG 0.5 mg (N=15) | NG 1 mg (N=14) | NG 2 mg (N=16) | SC Glucagon 1 mg (N=15)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pruritus (Eye disorders) | 0 (0) | 2 (2) | 2 (3) | 1 (1)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (6)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vessel puncture site haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vessel puncture site reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 2 (2) | 2 (2) | 2 (2) | 2 (2)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 4 (4) | 0 (0)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4) | 3 (3) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 4 (4) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days